CLINICAL TRIAL: NCT02981745
Title: Study of Safety, Efficacy and Pharmacokinetics of CT-1530 in Patients With Relapsed or Refractory B Cell Non-Hodgkin Lymphoma, Chronic Lymphocytic Leukemia, and Waldenstrom's Macroglobulinemia
Brief Title: Study of Safety,Efficacy and Pharmacokinetics of CT-1530 in Patients With Relapsed or Refractory B Cell Non-Hodgkin Lymphoma, Chronic Lymphocytic Leukemia, and Waldenstrom's Macroglobulinemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centaurus Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-1530-101
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Relapsed or Refractory B Cell Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Waldenstrom's Macroglobulinemia; Mantle Zone Lymphoma Refractory/Recurrent; Follicle Centre Lymphoma Diffuse; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT-1530 (Experimental)
  Interventions: Drug: CT-1530

INTERVENTIONS:
Drug: CT-1530 — Relapsed or Refractory B Cell Non-Hodgkin Lymphoma, Chronic Lymphocytic Leukemia, Waldenstrom's Macroglobulinemia, FL, Diffuse B-cell lymphoma, Mental-cell lymphoma

SUMMARY:
This is a phase I study of BTK inhibitor CT-1530 in patients with relapsed or refractory B cell non-Hodgkin lymphoma (B-NHL), chronic lymphocytic leukemia (CLL) or Waldenstrom's macroglobulinemia (WM).

The purpose of the study is to determine the MTD/RP2D of CT-1530, and evaluate its safety and tolerability as monotherapy in subjects with relapsed or refractory B cell non-Hodgkin lymphoma (B-NHL), chronic lymphocytic leukemia (CLL) or Waldenstrom's macroglobulinemia (WM).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of B cell Non-Hodgkin Lymphoma(according to World Health Organization [WHO] classification)including Chronic Lymphocytic Leukemia/Small cell Lymphocytic Leukemia (International Workshop),or Waldenstrom's Macroglobulinemia(Second International Workshop).
* Have failed ≥1 previous treatment for B-NHL/CLL/WM, and have relapsed or refractory disease following last prior treatment.
* Eastern Cooperative Oncology Group performance status of ≤ 1 and a life expectancy of at least 3 months.
* Measurable disease as per RECIST v1.1
* Availability of tumor sample
* Adequate hematologic function, as defined by neutrophils ≥ 1.0 x 10^9/L and platelets ≥ 50 x 10^9/L; patients with neutrophils < 1.0 x 10^9/L due to marrow infiltration are allowed to receive growth factors to bring pre-treatment neutrophils to ≥ 1.0 x 10^9/L.
* Adequate renal function, as defined by creatinine clearance of ≥ 50 ml/min (as estimated by the Cockcroft-Gault equation or as measured by nuclear medicine scan or 24 hour urine collection).
* Adequate liver function, as defined by AST and ALT ≤ 3 x ULN, and bilirubin ≤ 1.5 x ULN (unless documented Gilbert's syndrome).

Exclusion Criteria:

* Prior allogeneic bone marrow transplant
* Autologous stem cell transplant within 3 months of screening
* Active central nervous system involvement
* Subjects with autoimmune hemolytic anemia or immune thrombocytopenia
* Prior treatment with a Btk inhibitor
* Active uncontrolled infection
* History of malabsorption
* Uncontrolled illness, i.e cardiac, endocrine, respiratory, etc.
* History of myocardial infarction, acute coronary syndromes, coronary angioplasty and/or stenting with in the previous 6 months
* History of another currently active cancer
* History of major surgery within 4 weeks or minor surgery within 1 week
* Other medical or psychiatric illness or organ dysfunction
* HIV positive
* Positive for Hepatitis B surface antigen or Hepatitis C-virus

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of dose limiting toxicities (DLTs) during the first cycle of treatment (Phase I) | 28 days
  Maximum Tolerated Dose(s) (MTD(s)) and/or recommended phase 2 dose (RP2D(s)) of CT-1530 in Subjects With Relapsed or Refractory B Cell Non-Hodgkin Lymphoma, Chronic Lymphocytic Leukemia, Mental-cell lymphoma, Diffuse large B-cell lymphoma, FL and Waldenstrom's Macroglobulinemia

SECONDARY OUTCOMES:
Overall Response Rate (ORR) - Phase I | Up to 24 month
  Preliminary measure of anti-tumor activity of CT-1530
Progression free survival (PFS) per RECIST v1.1 - Phase I | Up to 24 months
  Preliminary measures of anti-tumor activity of CT-1530
Duration of response (DOR) | Up to 24 months
  Preliminary measure of anti-tumor activity of CT-707

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, M.D., Principal Investigator — Cancer Hospital of Chines Academy of Medical Sciences
Locations (1):
- Cancer Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No